CLINICAL TRIAL: NCT05939128
Title: A Multicentre, Single Arm, Non-interventional, Observational, Prospective Study to Assess the BRCA1/2m Prevalence, Treatment Approaches and Outcomes in HER2-negative High-risk Early Breast Cancer Patients in Russia
Brief Title: A Non-interventional Prospective Study of Early HER2-negative High-risk Breast Cancer and BRCA1/2 Mutations Prevalence in RussiA
Acronym: ERA
Status: Active, not recruiting | Type: Observational
Sponsor: AstraZeneca (Industry)
Responsible Party: Sponsor
Other Study IDs: D133HR00030
Record Dates: First submitted 2023-07-03; First posted 2023-07-11 (Actual); Last update posted 2026-02-12 (Actual); Status verified 2026-02

CONDITIONS: Breast Cancer
MeSH Terms: conditions — Breast Neoplasms

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Biospecimen Retention: Samples With DNA — tumor and blood samples

SUMMARY:
(Neo)adjuvant treatment approaches and outcomes

ELIGIBILITY:
Inclusion Criteria:

* Patients aged ≥ 18 years old

  -. Signed ICF, including patient's consent for genetic testing specimens from primary tumor and blood samples
* Early HER2-negative BC (stages 2 and 3)
* Compliance with at least 1 of the criteria for BRCA1/2 testing in accordance with the clinical guidelines of the Ministry of Health of the Russian Federation
* Unknown BRCAm status or negative BRCAm PCR test
* Performed surgical treatment (not more than 7 months before inclusion)

  -. High risk of recurrence according to one or more criteria:
  1. incomplete pathomorphological response (in case of neoadjuvant therapy)
  2. CPS-EG 3 scale score 3 and more (in case of neoadjuvant therapy)
  3. presence of ≥ 4 metastatic lymph nodes in HR+ pts (in case of only adjuvant therapy)
  4. ≥pT2 or ≥pN1 in TNBC pts (in case of only adjuvant therapy)
  5. Any other high risk criterion according to investigators opinion
* The presence of postoperative or biopsy FFPE

Exclusion Criteria:

* Participation in another clinical study with an investigational product during the last 3 months
* Confirmation that the subject was already included in this study before
* Absence of a written informed consent form; Data erroneously collected from subjects for which written consent is not available, will not be included in or will be deleted from the study database

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: Study population will consist of early breast cancer HER2-negative patients with high risk of recurrence with available medical history, surgery or biopsy FFPE from primary tumor. It is estimated that approximately 750 patients will be enrolled in approximately 25 sites
Sampling Method: Non-Probability Sample
Enrollment: 625 (Actual)
Dates: Start 2023-06-30 (Actual); Primary Completion 2027-09-30 (Estimated); Study Completion 2027-09-30 (Estimated)

PRIMARY OUTCOMES:
The primary objective of this study is to determine the prevalence of germline and somatic BRCA1/2 mutations in high-risk early HER2-negative breast cancer | 3 years
  The prevalence of germline and somatic BRCA1/2 mutations in high-risk early HER2-negative breast cancer will be presented as a number of missing and non-missing records, median, standard deviation, 95% confidence interval for median

SECONDARY OUTCOMES:
To describe treatment approaches of high-risk early HER2-negative breast cancer in routine practice in the general population, in the BRCAm and non-BRCAm population | 3 years
  Demographics, clinical characteristics, and treatment approaches will be summarized using descriptive statistics.
To determine invasive disease-free survival for high-risk early HER2-negative breast cancer in the general population, in the BRCAm and non-BRCAm population | 3 years
  The Kaplan-Meier method will be used to estimate the median (95% CI) IDFS and OS for the total sample and all subgroups. Cumulative survival curves will be created using Kaplan-Meier analysis
To determine 3-year OS for high-risk early HER2-negative breast cancer in the general population, in the BRCAm and non-BRCAm population | 3 years
  The Kaplan-Meier method will be used to estimate the median (95% CI) IDFS and OS for the total sample and all subgroups. Cumulative survival curves will be created using Kaplan-Meier analysis
To determine the prevalence of HRR mutations in HER2-negative breast cancer | 3 years
  Testing the archived tumour specimen and blood for BRCA1/2m and HRRm status
To determine invasive disease-free survival in the HRRm population (including BRCA1/2) | 3 years
  Testing the archived tumour specimen and blood for BRCA1/2m and HRRm status
To evaluate concordance between P53 expression and BRCAm | 3 years
  Testing the archived tumour specimen and blood
To assess the quality of life in patients with various types of adjuvant systemic therapy | 3 years
  completed WHOQOL-BREF questionnaire will be assessed

CONTACTS AND LOCATIONS:
Locations (19):
- Russia (19):
  - Research Site, Arkhangelsk
  - Research Site, Barnaul
  - Research Site, Belgorod
  - Research Site, Chelyabinsk
  - Research Site, Grozny
  - Research Site, Irkutsk
  - Research Site, Khanty-Mansiysk
  - Research Site, Krasnodar
  - Research Site, Krasnoyarsk
  - Research Site, Moscow
  - Research Site, Nal'chik
  - Research Site, Nyzhny Novgorod
  - Research Site, Ryazan
  - Research Site, Saint Petersburg
  - Research Site, Severodvinsk
  - Research Site, Sochi
  - Research Site, Ufa
  - Research Site, Vladivostok
  - Research Site, Yaroslavl